CLINICAL TRIAL: NCT03856138
Title: To Explore the Effect of Intestinal Microbiota and Fecal Inflammatory Marker on Childhood Gastroenteritis
Brief Title: Effect of Gut Microbiota and Fecal Inflammatory Marker on Childhood Gastroenteritis
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201507461B0
Record Dates: First submitted 2019-02-18; First posted 2019-02-27 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-01

CONDITIONS: Clinical Infection; Microbial Colonization; Gastroenteritis; Inflammatory Response; Probiotics
MeSH Terms: conditions — Communicable Diseases; Gastroenteritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bacteria DNA in feces of human
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- diarrhea with probiotics supplement: The children suffered from diarrhea, gastroenteritis oral probiotics during the clinical course
- diarrhea without probiotics supplement: The children suffered from diarrhea, gastroenteritis no oral probiotics during the clinical course
- healthy control: The children without diarrhea/ gastroenteritis

SUMMARY:
Childhood gastroenteritis establishes gastrointestinal disease and increase the economic burden, and the pediatric population is especially vulnerable to these gastrointestinal infections. The aim of this study is to evaluate the role of intestinal microbiota and their relationship with childhood gastroenteritis.

DETAILED DESCRIPTION:
Childhood gastroenteritis establishes gastrointestinal disease and increase the economic burden, and the pediatric population is especially vulnerable to these gastrointestinal infections. According to a World Health Organization report in 2003, the median incidence of diarrhea for all children age under 5 years was 3.2 episodes per child-year, and this number has not changed significantly since 1980s. In Taiwan, the enteric pathogens associated mortality is low, but the social burden and economic costs are substantial because of the high incidence.

Intestinal microflora are able to use the substances consumed in the diet: bacteria can transform complex polysaccharides and monosaccharides in short-chain fatty acids. Short-chain fatty acids are a source of energy for colonocytes and directly affect the storage of lipids and the absorption and metabolism of food, creating the so-called 'second meal effect'.

Qualitative and quantitative alterations of commensal flora may result in various gastrointestinal and extraintestinal diseases. One of the first interactions these bacteria have when interacting with the intestinal epithelial cells lining the GI tact.

The first aim of this study is to evaluate the role of intestinal microbiota and their relationship with childhood gastroenteritis. The second aim of this study is determining the inflammatory markers (such as fecal TNF-α, interleukin -6, calprotectin, lactoferrin) on the host of childhood gastroenteritis. The investigators try to seek to gain an advanced understanding effect of intestinal microbiota and fecal inflammatory marker in the childhood gastroenteritis.

ELIGIBILITY:
Inclusion Criteria:

* Children with or without diarrhea less than three days

Exclusion Criteria:

* diabetes
* chronic liver disease

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children with or without diarrhea less than three days, or healthy volunteers. The age of participants is from 6-month-old to 12-year-old.
Sampling Method: Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Fecal bacteria microbiota | the day of enrollment
  Bacteria count in feces
Fecal bacteria microbiota | 3 days after enrollment
  Bacteria count in feces
Fecal bacteria microbiota | 7 days after enrollment
  Bacteria count in feces
Fecal bacteria microbiota | 1 month after enrollment
  Bacteria count in feces

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Chang Chen, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided